CLINICAL TRIAL: NCT05243966
Title: Registry of Myriad™ Utilization in Soft Tissue Reconstruction Procedures
Brief Title: Myriad™ Augmented Soft Tissue Reconstruction Registry
Acronym: MASTRR
Status: Recruiting | Type: Observational
Sponsor: Aroa Biosurgery Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP.SUR.001
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Wound Dehiscence; Necrotizing Soft Tissue Infection; Lower Extremity Wound; Pilonidal Sinus; Anal Fistula; Hidradenitis Suppurativa; Pressure Injury
Keywords: Soft tissue reconstruction; Limb salvage; Extracellular matrix; Soft tissue reinforcement; Wound reconstruction; Regenerative medicine
MeSH Terms: conditions — Pilonidal Sinus; Rectal Fistula; Hidradenitis Suppurativa; Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Myriad™: Ovine forestomach matrix sheet graft and morselized extracellular matrix
  Interventions: Device: Myriad Matrix™ and Myriad Morcells™

INTERVENTIONS:
Device: Myriad Matrix™ and Myriad Morcells™ — Ovine forestomach matrix sheet graft and morselized extracellular matrix

SUMMARY:
This is an observational study designed to evaluate the safety and clinical outcomes of Myriad™ in soft tissue reconstruction procedures. The study will enroll participants who are undergoing a surgical procedure, where the attending physician will use Myriad™ as part of the surgical intervention.

DETAILED DESCRIPTION:
This is an observational, multi-center, single arm, Phase IV study, designed to evaluate the safety and clinical outcomes of Matrix and Morcells in soft tissue reconstruction procedures.

The study is a registry study and will enroll participants who are undergoing a surgical procedure, and where the attending physician will use Myriad Matrix™ and/or Morcells™ as part of the surgical intervention.

Participants enrolled in the study will be undergoing a range of surgical procedures involving the reconstruction of soft tissues, including but not limited to:

* Abdominal dehiscence
* Necrotizing soft tissue infection (NSTI)
* Lower extremity complex non-healing wounds (limb salvage)
* Pilonidal sinus disease
* Anal fistula
* Hidradenitis suppurativa reconstruction
* Pressure injury reconstruction

Other procedure types may be included at the discretion of the Investigator/Research Team.

Participants that are being enrolled in the study would otherwise be undergoing their surgical procedure with either of the Myriad™ devices as part of Standard of Care (SoC).

The pre-operative care and preparation of the surgical site (prior to the application of Myriad™ devices) shall be undertaken at the discretion of the attending physician and per their institutional protocols and procedures. Surgical technique for the participants reconstruction is at the discretion of the attending physician. Use of Myriad Matrix™ or Morcells as part of the surgery shall be per the products Instructions for Use. Myriad Matrix™ devices may be implanted or used for dermal regeneration as part of the participants surgical procedure. Myriad Morcells™ may be used for dermal regeneration and in combination with the Myriad Matrix™ devices. The participants post-operative care is at the discretion of the attending physician.

Early and late-stage healing outcomes will be assessed as part of the study and as part of standard of care.

Through the course of treatment and following up care de-identified patient data (quantitative qualitative assessment measures and digital images) will be captured and from the basis of the registry dataset.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and to comply with the requirements of Clinical Investigational Plan
* Male or female patients aged 18 years or above
* Patients where Matrix and/or Morcells were used as part of their soft tissue reconstruction procedure
* Subject that are willing and able to comply with all aspects of the treatment and evaluation schedule

Exclusion Criteria:

* Patients with known sensitivity to ovine (sheep) derived material
* Patients with full thickness ('third degree') burns
* Patients with wounds with uncontrolled clinical infection (CDC Contamination Grade=4)
* Any medical condition or serious intercurrent illness that, in the opinion of the investigator, may make it undesirable for the patient to participate in the study
* Patient is currently participating or has participated in another clinical study within past 30 days prior to enrollment
* Pregnant or lactating women
* Any subject who, at the discretion of the Investigator, is not suitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is being carried out at approximately 10 sites in the U.S. Across all sites, about 300 individuals will participate in the study where the Investigator is planning to utilize Myriad™ as a part of their surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment emergent adverse events during the study | 3 years
  Nature, frequency, and severity of adverse events

SECONDARY OUTCOMES:
Time (weeks) to complete healing | Up to 52 weeks
  When Myriad™ is used in soft tissue reinforcement the time to would closure will be recorded
Percentage of surgical complications | Up to 3 months
  Reporting the incidence of infection, seroma/hematoma, dehiscence from surgical procedures
Time (weeks) to 100% granulation | Up to 3 months
  Where applicable, when Myriad™ is used for dermal regeneration, the time until full graft integration will be recorded
Percentage of split thickness skin graft take at 1 week post Matrix™ application | 1 week post application
  Where applicable, when Myriad™ is used for dermal regeneration and a split thickness skin graft is used the percentage of graft take at 1 week will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Tracee Short, MD, Study Chair — Short Consulting Group, LLC
Locations (12):
- United States (12):
  - Surgery Group LA, Los Angeles, California
  - Associates in Medicine & Surgery, Fort Myers, Florida
  - Asencion Sacred Heart, Pensacola, Florida
  - Northeast Georgia Medical Center, Inc., Gainesville, Georgia
  - University Medical Center, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Nuvance Health Vassar Brothers Medical Center, Poughkeepsie, New York
  - Moses H Cone Memorial Hospital Operating Corporation, Greensboro, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Tower Health Reading Hospital, West Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided